CLINICAL TRIAL: NCT03104634
Title: The Effects of Inhaled Aclidinium Bromide/Formoterol Fumarate on Inspiratory Pleural Pressures in Smokers: a Randomized, Double-blind, Placebo-controlled, Cross-over Trial
Brief Title: The Effects of Inhaled Aclidinium Bromide/Formoterol Fumarate on Inspiratory Pleural Pressures in Smokers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Benjamin McDonald Smith, Assistant professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-2748
Record Dates: First submitted 2017-03-29; First posted 2017-04-07 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — aclidinium bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Matched placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active arm (Experimental): Aclidinium bromide/formoterol fumarate dihydrate 400 mcg/12 mcg Twice daily (once in the morning, once in the evening) 7-days
  Interventions: Drug: Aclidinium bromide/formoterol fumarate dihydrate
- Placebo arm (Placebo Comparator): Placebo Twice daily (once in the morning, once in the evening) 7-days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aclidinium bromide/formoterol fumarate dihydrate — Cross-over design with washout interval. Randomized order of active and placebo arm
  Other Names: DUAKLIR™ GENUAIR®
  Arms: Active arm
Drug: Placebo — Placebo and delivery device matched to active intervention
  Arms: Placebo arm

SUMMARY:
This short-term study aims to prove the potential cardio-protective physiological effect of inhaled aclidinium bromide/formoterol fumarate on inspiratory pleural pressures.

Smoking is associated with gas-trapping (hyperinflation), even in the absence of chronic obstructive pulmonary disease. Breathing in the presence of gas-trapping requires large negative inspiratory pleural pressures, which are transmitted to the surface of the heart and increase cardiac wall stress.

Inhaled aclidinium bromide and formoterol fumarate has been shown to reduce gas-trapping, but the impact on inspiratory pleural pressures and biomarkers of cardiac stress in smokers is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Current and former smokers with ≥20 pack-years of smoking history
* Gas-trapping (residual volume >110% predicted)

Exclusion Criteria:

Physician-diagnosis of chronic obstructive pulmonary disease in the past 1 year and regular use of long-acting antimuscarinic (LAMA) and/or long-acting beta-agonist (LABA) (i.e., at least 30 consecutive days)

* Physician-diagnosis of asthma in the past 5 years
* Regular inhaled corticosteroid (ICS) use in the past 5 years (i.e., at least 30 consecutive days)
* Physician-diagnosis of other lung diseases (sarcoidosis, tuberculosis, cystic fibrosis, pulmonary fibrosis, lung cancer), or long-term oxygen therapy
* Respiratory tract infection within 4-weeks
* Physician-diagnosis of arrhythmia, or significant valvular disease.
* Physician-diagnosis of myocardial infarction, unstable angina or heart failure requiring unscheduled outpatient or emergency department visit within 6-months.
* Arrhythmia or prolonged corrected QT (QTc) on electrocardiogram.
* Inability to use study inhaler
* Glaucoma
* Benign prostatic hypertrophy
* Pregnancy
* Allergy to the study treatment, salbutamol, lidocaine, or severe milk protein allergy (note: lactose intolerance is not an exclusion criteria)
* Contraindications to anti-cholinergic, beta-agonist, or cardiopulmonary exercise testing with manometry
* Inability to provide written informed consent

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-reported gender
Enrollment: 43 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Inspiratory pleural pressures at rest and throughout incremental exercise (cmH2O) | After 7-days of active or placebo drug
  Mean difference in inspiratory pleural pressure measured by esophageal manometry at rest and throughout incremental exercise

SECONDARY OUTCOMES:
Resting and exercise-induced changes in plasma natriuretic peptide concentrations (plasma concentration) | After 7-days of active or placebo drug
  Mean difference in atrial natriuretic peptide (exercise induced-changes) and n-terminal pro-B-type natriuretic peptide (resting).
Resting and dynamic lung volumes (end-inspiratory/end-expiratory lung volume) | After 7-days of active or placebo drug
  Static and operating lung volumes
Effect modification by gender (self-reported). | After 7-days of active or placebo drug
  Interaction term added to regression model for gender.
Effect modification by smoking status (self-reported). | After 7-days of active or placebo drug
  Interaction term added to regression model for smoking status.
Effect modification by hypertension status (Joint National Committee criteria). | After 7-days of active or placebo drug
  Interaction term added to regression model for hypertension status.
Effect modification by hyperinflation severity (Residual lung volume). | After 7-days of active or placebo drug
  Interaction term added to regression model for hyperinflation severity.
Effect modification by spirometric chronic obstructive pulmonary disease (COPD) status (forced expired volume in 1 second-to-forced vital capacity ratio below 0.7). | After 7-days of active or placebo drug
  Interaction term added to regression model for spirometric COPD status.

CONTACTS AND LOCATIONS:
Overall Officials: B M Smith, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre Research Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided